CLINICAL TRIAL: NCT03265925
Title: Brain Network Activation Analysis in Epilepsy
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM-40
Record Dates: First submitted 2017-08-20; First posted 2017-08-29 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Epilepsy; Epilepsy, Temporal Lobe
MeSH Terms: conditions — Epilepsy; Epilepsy, Temporal Lobe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Epilepsy patients Right Temporal Lobe: Epilepsy patients with seizures originating from the right temporal lobe
- Epilepsy patients Left Temporal Lobe: Epilepsy patients with seizures originating from the left temporal lobe
- Healthy: Healthy controls

SUMMARY:
This is a prospective study investigating the utility of Brain Network Activation (BNA) analysis in patients with epilepsy.

DETAILED DESCRIPTION:
BNA technology is based on a network model to depict functional connectivity. The descriptive network model approach provides insights regarding inter-connectivity of brain networks and can describe the temporal-spatial brain activation patterns applied to various types of data-sets including EEG, MEG and fMRI.

In this study it is proposed that synchronization in brain activity may be disrupted in patients who experience frequent seizures and may correspond to functional impairments (e.g., memory, processing speed). As such, BNA analysis may provide additional data that complement current functional assessments, inform clinical assessment and management of epilepsy, and identify subgroups of patients that might be at risk for poor treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be between ages 18-50 years old
* Able to speak, read and understand English sufficiently to understand the nature of the study, and to allow completion of all study assessments
* Willingness to participate and able to give informed consent
* If corrected vision: only Glasses should be used during the study testing

Exclusion Criteria:

* History of significant head trauma
* Evidence of other neurologic disease
* Any diagnosed psychiatric or systemic condition that could lead to a change in brain activity or volume (e.g., stroke, Alzheimer's disease, alcoholism).
* Currently with lice or open wounds on scalp
* Significant sensory deficits
* Use of a hearing aid that occupies the ear canal
* Substance abuse in the last 3 months and any clinically significant substance dependency
* Additional exclusion criteria for controls are a history of any neurological disease or psychological illness.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from the long-term EEG monitoring floor and outpatient EEG laboratory. Controls will be recruited in response to advertisements. All participants will be given the BNA Auditory Go/NoGo task. Patient identity will be coded with a master record kept on a password protected computer in the laboratory. Deidentified data will be sent to ElMindA for scoring of the BNA test. Patient data from electronic medical records will be extracted along with patient MRI data processed.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Assess the BNA database for Epilepsy population and healthy controls. | Epilepsy subjects will perform the BNA testing at baseline prior to change in medication if applicable and 3-10 days following change in medication when applicable.
  Functional networks of brain activity in Epilepsy (Right and Left lobe) and healthy control individuals measured using analysis of EEG Event Related Potential (ERP) data. Clinical assessments battery will be utilized in order to examine different sets of BNA database for Epilepsy pathology and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Travis Stoub, PhD, Principal Investigator
Locations (1):
- RUSH University medical center, Chicago, Illinois, United States